CLINICAL TRIAL: NCT04586322
Title: Association Between Erosive Tooth Wear Progression and Dietary Risk Factors in Chileans Adolescents.
Brief Title: Association Between Erosive Tooth Wear Progression and Dietary Risk Factors.
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2809ErosionC
Record Dates: First submitted 2020-09-28; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Tooth Erosion; Tooth Wear; Erosion; Dental Erosion
Keywords: Tooth Erosion; Tooth wear
MeSH Terms: conditions — Tooth Erosion; Tooth Wear | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention, (observational study). — From every participant the following information was recorded for further analysis:
  * BEWE score- Basic erosive tooth wear examination (from 2 calibrated examiners) to diagnose the presence of erosive tooth wear.
  * Their answer to a validated questionnaire assessing the dietary habits based in the frequency of acidic diet.
  * 2 Intra oral scans (IOS): Baseline and follow up (1 year after baseline) to perform a quantification of tissue loss (in Volume loss per mm3) using Wearcompare software.

SUMMARY:
Study to determine if whether or not exist an association between the tissue loss (ETW progression) and the frequency of an acidic diet. To accomplish the aim, a quantitative analysis of intraoral scans of study models will be performed to identify erosive tooth wear progression in a group of Chilean adolescents.

First, participants with different intake of dietary acids will be compared in terms of their baseline sociodemographic and clinical characteristics. Second, the association between baseline frequency of dietary acids and changes in volume loss over time will be evaluated using linear mixed models to account for the data structure (repeated assessments nested within teeth and teeth nested within children). Models will be adjusted for demographic factors, family socioeconomic position, health behaviours and chronic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male and female (age range 10-18) assisting in a school with low socioeconomic status.

They must have: -Complete record of questionnaires

* Baseline and Follow-up Intra oral scanners (with correct alignment when using Wearcompare software)
* BEWE scores
* Signed Inform consent

Exclusion Criteria:

* Patients not willing to participate
* Patients wearing orthodontic appliances

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents subscribed at 2 Chilean high schools of the Community La Pintana, Santiago de Chile (Colegio Nocedal and Colegio Almendral). Schools belong to a low socio economic status sector.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Volume loss | 14 months
  Volume Loss in mm3 in patients having a frequent consumption of dietary acids (cut off to decide) Volume loss will be determined by aligning the marker teeth of each participant: 1.1-2.1-1.6-2.6-3.6 and 4.6.

SECONDARY OUTCOMES:
Dietary Risk factors | 14 months
  Frequency of consumption of dietary acids (Possible cut off: > 1 a day)

CONTACTS AND LOCATIONS:
Locations (1):
- Francisca Marro, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No